CLINICAL TRIAL: NCT03512626
Title: Clinical Evaluation of Multifocal Intraocular Lens: OPTIVIS.TM (Evolución clínica de Lente Intraocular Multifocal: OPTIVIS.TM)
Brief Title: Clinical Evaluation of Multifocal Intraocular Lens: OPTIVIS.TM
Acronym: MFIOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, ANNA MARTÍNEZ PALMER, Head of Ophthalmology Department, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/5432/I
Record Dates: First submitted 2018-04-08; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Cataract Senile; Lenses, Intraocular
Keywords: OptiVis; hybrid multifocal intraocular lens; multifocal intraocular lens; presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Consecutive patients with bilateral cataract were included after meeting all the inclusion and none of exclusion criteria and when written informed consent was obtained from all patients.
  Patients were randomly assigned to have bilateral implantation with either a monofocal IOL (AR40e, AMO-Abbot 30 Laboratories Inc. Abbot Park, Illinois, USA) or multifocal IOL (OptiVis™, Aaren Scientific, Inc, Ontario, CA, USA).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multifocal IOL (OptiVis) (Experimental): Ambulatory surgery was performed by the same, experienced surgeon, under topical anesthesia, using as a technique phacoemulsification with small incision (2.75) in clear cornea in the most curved meridian.
  The randomly assigned IOL (in this arm: a hybrid (refractive-diffractive) multifocal IOL (OptiVis, Aaren Scientific) was implanted in the capsular bag. The second eye with the same type of lens of the first eye was operated within 2-4 weeks.
  Interventions: Device: OptiVis, Aaren Scientific
- Monofocal IOL (Active Comparator): Ambulatory surgery was performed by the same, experienced surgeon, under topical anesthesia, using as a technique phacoemulsification with small incision (2.75) in clear cornea in the most curved meridian.
  The randomly assigned IOL (in this arm: a monofocal IOL (AR40e, AMO) was implanted in the capsular bag. The second eye with the same type of lens of the first eye was operated within 2-4 weeks.
  Interventions: Device: Monofocal IOL

INTERVENTIONS:
Device: OptiVis, Aaren Scientific — All the surgeries were performed under topical anesthesia using a standard phacoemulsification procedure with Infiniti Vision System (all from Alcon Laboratories, Inc, Fort Worth, TX).
  Other Names: a hybrid multifocal intraocular lens
  Arms: Multifocal IOL (OptiVis)
Device: Monofocal IOL — All the surgeries were performed under topical anesthesia using a standard phacoemulsification procedure with Infiniti Vision System (all from Alcon Laboratories, Inc, Fort Worth, TX).
  Other Names: AR40e, AMO-Abbot 30 Laboratories Inc.
  Arms: Monofocal IOL

SUMMARY:
This study evaluated visual outcome after cataract surgery with bilateral implantation of either a diffractive - refractive (hybrid) multifocal intraocular lens (MFIOL) or monofocal intraocular lens (IOL) as a control grup.

DETAILED DESCRIPTION:
PURPOSE: To present the outcomes of hybrid multifocal and monofocal intraocular lenses (IOL)

SETTING: Parc de Salut Mar, Universidad Pompeu-Fabra - Autónoma, Barcelona, Spain.

DESIGN: Prospective clinical trial.

METHODS: Consecutive patients with bilateral cataract were included. Phacoemulsification with randomized implantation of either a monofocal IOL (AR40e, AMO-Abbot 30 Laboratories Inc. Abbot Park, Illinois, USA) or multifocal IOL (OptiVis™, Aaren Scientific, Inc, Ontario, CA, USA) was performed by the same surgeon and under the same conditions. Over a 3-month follow-up, the main outcome measures were uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), uncorrected intermediate visual acuity at 60 cm (UIVA), distance-corrected intermediate visual acuity (DCIVA), uncorrected near visual acuity at 33 cm (UNVA), distance-corrected near visual acuity (DCNVA), spherical equivalent (SE), contrast sensitivity (CS), presence of dysphotopsia, use of spectacles and patient satisfaction with the test VF-14 (Visual Function Index) .

ELIGIBILITY:
Inclusion Criteria:

* senile cataract with Snellen visual acuity ≤ 0.5,
* motivation for spectacle independence for near vision (as the study was conducted in Spanish public health care system, entering study was the only option to get multifocal lens, as they are not provided by public health care, and the patients were conscious of the possibility of randomization to monofocal group.)

Exclusion Criteria:

* corneal astigmatism ≥ 1.10 diopters (D) and irregular astigmatism,
* axial length < 21.5 or ≥ 25 mm,
* pupillary diameter in mesopic conditions in distance vision ≤ 2.5 mm and ≥ 6 mm,
* ocular pathology that could affect the visual function and/or intraocular lens centering and intraoperative or postoperative complications.
* highly demanding patients and those whose profession could be affected by a multifocal design (professional drivers, jewelers etc.) were also excluded (as in the Spanish public health care system secondary procedures needed to satisfy patients' expectation, such as LRI´s, LASIK, PRK´s, are not available).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

PRIMARY OUTCOMES:
Visual function | The last follow-up visit (3 months after the surgery)
  Changes in visual acuity in logMAR: uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA) at 6 m, uncorrected intermediate visual acuity (UIVA), distance-corrected intermediate visual acuity (DCIVA) at 60 cm (in the OptiVis group only, as they were supposed to provide intermediate distance vision in contrary to monofocal lenses), uncorrected near visual acuity (UNVA) and distance-corrected near visual acuity (DCNVA) at 33 cm. All measured using Snellen acuity charts under photopic conditions.

SECONDARY OUTCOMES:
Contrast sensitivity (CS) | The last follow-up visit (3 months after the surgery)
  Changes in monocular and binocular CS were measured in mesopic conditions, without glare at spatial frequencies of 1.5, 3, 6, 12 and 18 cycles per degree (cpd) using the Functional Acuity Contrast Test (FACT, OPTEC 6500®, Stereo Optical Co. Inc)
Refractive Outcomes | The last follow-up visit (3 months after the surgery)
  The predictability of the refractive outcome. Postoperative spherical equivalent (SE) and SE within ±0.50 D of the attempted spherical correction (emmetropy) and within ±1.00 D of the attempted spherical correction (emmetropy).
Spectacle dependence | The last follow-up visit (3 months after the surgery)
  Spectacle dependence, determined by questionnaire (Do you wear glasses for distance/near vision?).
Presence of dysphotopsia | The last follow-up visit (3 months after the surgery)
  Presence of dysphotopsia (halos, glare), spontaneously mentioned or elicited in response to questioning were determined by questionnaire.
Patient satisfaction | The last follow-up visit (3 months after the surgery)
  Patient satisfaction was also assessed with the VF-14 test, consisting of 14 questions evaluating various patient activities.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Martinez Palmer, PhD, Principal Investigator — Parc de Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data are available now as the conducted study was finished and until the publication will be in press. After that all data will be available via journal requests
Access Criteria: Requesters will be required to sign a Data Access Agreement

REFERENCES:
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Cochener B, Lafuma A, Khoshnood B, Courouve L, Berdeaux G. Comparison of outcomes with multifocal intraocular lenses: a meta-analysis. Clin Ophthalmol. 2011 Jan 7;5:45-56. doi: 10.2147/OPTH.S14325. PMID 21311656
- [Background] Piovella M, Bosc JM. Clinical evaluation of the OptiVis multifocal intraocular lens. Adv Ther. 2011 Nov;28(11):1012-20. doi: 10.1007/s12325-011-0064-7. Epub 2011 Oct 31. PMID 22057725
- [Background] Calladine D, Evans JR, Shah S, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD003169. doi: 10.1002/14651858.CD003169.pub3. PMID 22972061
- [Background] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Derived] Dyrda A, Martinez-Palmer A, Martin-Moral D, Rey A, Morilla A, Castilla-Marti M, Arones-Santivanez J. Clinical Results of Diffractive, Refractive, Hybrid Multifocal, and Monofocal Intraocular Lenses. J Ophthalmol. 2018 Jun 25;2018:8285637. doi: 10.1155/2018/8285637. eCollection 2018. PMID 30046464